CLINICAL TRIAL: NCT06174987
Title: A Master Rollover Study to Provide Continued Access to and Assess Long-Term Safety of the Study Drug(s)
Brief Title: A Study to Provide Continued Access to and Assess Long-Term Safety of the Study Drug(s)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROMast-001; 2023-506330-73-00 (Other: EU CTIS)
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Advanced Cancer; Metastatic Cancer
Keywords: Advanced cancer; Metastatic cancer; T-DXd; DS8201a
MeSH Terms: conditions — Neoplasm Metastasis | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- T-DXd (Experimental): Participants who choose to continue treatment with T-DXd may be enrolled. Participants who were on the comparator arm in the parent study will be provided the option to access the drug through standard of care (SoC) or other available options.
  Participants will remain on their current dosage regimen of T-DXd as the last dose administered in the parent study, unless they experience an AE that requires dose reduction at the EOT of the parent study, in which case the starting dose in this study will be the next lower dose-level.
  Interventions: Drug: T-DXd

INTERVENTIONS:
Drug: T-DXd — T-DXd (DS8201a) will be administered as an intravenous (IV) infusion, on Day 1 of each 21-day cycle according to the dosage regimens
  Other Names: DS8201a

SUMMARY:
This open-label, multicenter, rollover study will provide continued treatment for participants deriving benefit from different therapies received in studies sponsored by Daiichi Sankyo, Inc. (DS) or DS/Astra Zeneca (AZ)-sponsored study (eg. DS8201-A-J101, DS8201-A-U201, DS8201-A-U204, DS8201-A-U207, DS8201-A-U303).

DETAILED DESCRIPTION:
This Master Rollover Study includes sub-protocols with different study drugs. This Master Rollover Protocol describes core study elements that are applicable to all study drugs that will be provided under the Rollover Study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form, prior to the start of any study-specific qualification procedures and willing to comply with all study requirements.
* Currently enrolled in a DS or DS/AZ-sponsored parent study that has met EOS definition.
* No evidence of progressive disease and determined to have investigator-assessed clinical benefit from continued treatment with a DS or DS/AZ alliance study drug(s).

Exclusion Criteria:

* Participants with any unresolved/ongoing AE(s) that meets the study drug discontinuation criteria
* Participant who has been off T-DXd therapy for >18 weeks (126 days) between the last dose from the parent study and the initiation of study drug administration on this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2026-08-03 (Estimated); Study Completion 2028-01-17 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Reporting Treatment-emergent Adverse Events Leading to Study Drug discontinuation and/or Dose Reduction, Treatment-emergent Serious Adverse Events (TESAEs), and Treatment-emergent Adverse Events of Special Interest (AESIs) | Baseline until disease progression, loss of clinical benefit, death, adverse event, pregnancy, withdrawal of consent, access to commercial supply, physician decision, or study closure, whichever occurs first, up to approximately 2 years 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (28):
- United States (2):
  - Miami Cancer Institute, Miami, Florida
  - Duke University - Trent Center, Durham, North Carolina
- Australia (2):
  - Flinders Medical Center, Bedford Park
  - Monash Medical Center, Melbourne
- Grand Hôpital de Charleroi, Charleroi, Belgium
- Brazil (3):
  - Instituto Aericas, Rio de Janeiro
  - A.C. Camargo Cancer Center, São Paulo
  - IBCC Nucleo de Pequisa e Ensino, São Paulo
- Institut Gustave Roussy, Villejuif, France
- Rabin Medical Center, Petah Tikva, Israel
- Italy (2):
  - Ospedale San Raffaele, Milan
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
- National Cancer Center Hospital, Chūō, Japan
- South Korea (7):
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Jongno-gu
  - Severance Hospital, Yonsei University, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitari Dexeus, Distrito de Les Corts
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital Ruber Internacional, Madrid
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Royal Surrey County Hospital, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/